CLINICAL TRIAL: NCT06941714
Title: Evaluating the Effects of Cognitive Load on Postural Stability and Balance Recovery Mechanisms in Younger Adults
Brief Title: Cognitive Load Effects on Balance and Postural Stability in Young Adults
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Health Services Research
Other Study IDs: REC/02023 Imran Amjad
Record Dates: First submitted 2025-04-07; First posted 2025-04-24 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: Balance; Cognitive Load
Keywords: Performance

STUDY DESIGN:
Intervention Model Description: Research
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Baseline Balance Assessment (No Intervention): All participants who fall in the eligibility criteria will stand on force plates to check the static balance.
- Static Balance along with Cognitive Loading (Experimental): All participants who fall in the eligibility criteria will stand on force plates to check static balance and undergo two different types of cognitive loading
  Interventions: Other: Working Memory Task; Other: Visual and Verbal Fluency Task
- Perturbation (Experimental): All participants who fall in the eligibility criteria will stand on force plate and perturbation is given to check balance recovery.
  Interventions: Other: Perturbation
- Perturbation along with Cognitive Loading (Experimental): All participants who fall in the eligibility criteria will stand on force plate and perturbation is given to check balance recovery and undergo two different types of cognitive loading.
  Interventions: Other: Perturbation; Other: Working Memory Task; Other: Visual and Verbal Fluency Task

INTERVENTIONS:
Other: Perturbation — Jack is attached to force plates and it is used to give perturbation when participants are standing on force platform. Balance is assessed after perturbation and readings will be taken through HRV and GSR.
  Arms: Perturbation; Perturbation along with Cognitive Loading
Other: Working Memory Task — Arithmetic test (Backward counting with serial 3 subtraction and articulation): participants are asked to count out loud backward with serial subtraction of 3 from each number, starting with a random number provided by the researcher. while participants are standing on force plates. During all this process cognitive loading will be measured through Heart Rate Variability (HRV) and Galvanic Skin Response (GSR).
  Arms: Perturbation along with Cognitive Loading; Static Balance along with Cognitive Loading
Other: Visual and Verbal Fluency Task — Modified Stroop test or Stroop color word test: Participants are asked to name the color of ink that each word is printed. The test will appear on screen while participants are standing on force plates. During all this process cognitive loading will be measured through Heart Rate Variability (HRV) and Galvanic Skin Response (GSR).
  Arms: Perturbation along with Cognitive Loading; Static Balance along with Cognitive Loading

SUMMARY:
* The aim is to determine the impact of cognitive load on balance recovery mechanisms following perturbations in young adults.
* To evaluate how secondary task is influenced by cognitive load and vice versa.
* To compare the impact of cognitive load on balance recovery mechanisms following perturbations in male and female young adults.
* This study interrelates the cognitive load, postural stability, balance recovery in the result of perturbation and effects on participants.

DETAILED DESCRIPTION:
Maintaining balance is an important skill that requires coordination and is crucial for human beings. The Central Nervous System (CNS) plays an important role in maintaining balance, postural stability, and postural correction in response to sudden perturbation. The subcortical brain region contributes to balance maintenance and postural stability is regulated by the cerebral cortex. Balance is defined as the "Body's ability to keep its center of gravity within the base of support either standing or walking". On a regular basis people encounter perturbations (traveling on a bus while standing) that challenge balance, to overcome unexpected perturbations there must be activation of postural muscles to maintain the center of gravity within the base of support and prevent fall. Individuals mostly use ankle strategy or hip strategy to recover from perturbation and prevent fall. Anticipatory postural adjustment is a critical component of postural stability. recently cognition and postural control have received attention, there are studies that claim that dual-task design has been used to show the relation between posture and cognitive functioning. In the dual-task paradigm two tasks are performed simultaneously to divert the attention of an individual to an external source (counting backward etc.) while performing another task. Divided attention is commonly required in daily life while performing dual tasking and multitasking activities, if attention is not properly divided among task it will results in decline in performance which causes impairment of balance and fall.To prevent this, balance must be recovered from perturbation. The purpose is to assess effect of cognitive loading and recovery from perturbations along with balance maintenance and fulfillment of research gap that study should be performed with multiple methods of cognitive loading. That's why different methods for cognitive loading are used in current study which shows that how varying levels of cognitive load influence postural stability and balance in dual-task conditions. This research can help in rehabilitation programs in which specific interventional designs and treatment protocols are made to improve balance under the influence of cognitive load. Provide awareness to people on a societal level to improve their balance and posture maintenance under a mental workload.

ELIGIBILITY:
Inclusion Criteria

* Participants between age of 18 to 30 (university Students)
* Sufficient physical function to stand independently.
* Self-reported independent ambulation.
* Participant willingness to participate.

Exclusion Criteria:

* History of neurological or vestibular disorders.
* Self-reported presence of musculoskeletal condition.
* Disorders of spine, pelvic girdle and lower limb.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — All male and female healthy students are eligible to participate.
Enrollment: 80 (Estimated)
Dates: Start 2025-04-23 (Actual); Primary Completion 2025-07-30 (Estimated); Study Completion 2025-07-30 (Estimated)

PRIMARY OUTCOMES:
Centre of Pressure | Baseline
  Force plates are used to measure data quantitatively and analyze postural stability through the displacement of COP from forces and moments. A force platform is used in conditions when the force platform is not moving (static posturography) and when the force platform is moving (dynamic posturography). It has the capability of measuring ground reaction forces in three directions and the moment of force. Each of the platforms was connected to a dedicated computer with relevant software and valid controllers.
Centre of Pressure (2nd reading) | Periprocedural
  Force plates are used to measure data quantitatively and analyze postural stability through the displacement of COP from forces and moments. A force platform is used in conditions when the force platform is not moving (static posturography) and when the force platform is moving (dynamic posturography). It has the capability of measuring ground reaction forces in three directions and the moment of force. Each of the platforms was connected to a dedicated computer with relevant software and valid controllers.
  2nd reading will be taken to measure static balance along with cognitive loading.
Centre of Pressure (3rd reading) | Periprocedural
  Force plates are used to measure data quantitatively and analyze postural stability through the displacement of COP from forces and moments. A force platform is used in conditions when the force platform is not moving (static posturography) and when the force platform is moving (dynamic posturography). It has the capability of measuring ground reaction forces in three directions and the moment of force. Each of the platforms was connected to a dedicated computer with relevant software and valid controllers.
  3rd reading will be taken at the time of perturbation without cognitive loading.
Centre of Pressure (4rth reading) | Periprocedural
  Force plates are used to measure data quantitatively and analyze postural stability through the displacement of COP from forces and moments. A force platform is used in conditions when the force platform is not moving (static posturography) and when the force platform is moving (dynamic posturography). It has the capability of measuring ground reaction forces in three directions and the moment of force. Each of the platforms was connected to a dedicated computer with relevant software and valid controllers.
  4rth reading will be taken at the time of perturbation along with cognitive loading.
Postural Sway | Baseline
  It is assessed through a force plate when the subject is standing on it.
Postural Sway (2nd reading) | Periprocedural
  It is assessed through a force plate when the subject is standing on it. 2nd reading will be taken to measure static balance along with cognitive loading.
Postural Sway (3rd reading) | Periprocedural
  It is assessed through a force plate when the subject is standing on it. 3rd reading will be taken at the time of perturbation without cognitive loading.
Postural Sway (4rth reading) | Periprocedural
  It is assessed through a force plate when the subject is standing on it. 4rth reading will be taken at the time of perturbation along with cognitive loading.
Balance Recovery | Periprocedural
  Jack is attached to force plates, and it is used to give a perturbation when the participant is standing on the force platform, and balance is assessed after the participant recovers from the perturbation. 1st reading will be taken to measure static balance without cognitive loading.
Balance Recovery (2nd reading) | Periprocedural
  Jack is attached to force plates, and it is used to give a perturbation when the participant is standing on the force platform, and balance is assessed after the participant recovers from the perturbation. 2nd reading will be taken to measure static balance along with cognitive loading.
Heart Rate Variability | Baseline
  Heart Rate Variability is a beat-to-beat fluctuation in normal sinus rhythm, and it arises due to variation between the sympathetic and parasympathetic divisions of the autonomic nervous system. Heart Rate Variability (HRV) is measured by using ECG signals. There is a positive association between HRV indices and cognitive performance.
Heart Rate Variability (2nd reading) | Periprocedural
  Heart Rate Variability is a beat-to-beat fluctuation in normal sinus rhythm, and it arises due to variation between the sympathetic and parasympathetic divisions of the autonomic nervous system. Heart Rate Variability (HRV) is measured by using ECG signals. There is a positive association between HRV indices and cognitive performance. 2nd reading will be taken to measure static balance along with cognitive loading.
Heart Rate Variability (3rd reading) | Periprocedural
  Heart Rate Variability is a beat-to-beat fluctuation in normal sinus rhythm, and it arises due to variation between the sympathetic and parasympathetic divisions of the autonomic nervous system. Heart Rate Variability (HRV) is measured by using ECG signals. There is a positive association between HRV indices and cognitive performance. 3rd reading will be taken at the time of perturbation without cognitive loading.
Heart Rate Variability (4rth reading) | Periprocedural
  Heart Rate Variability is a beat-to-beat fluctuation in normal sinus rhythm, and it arises due to variation between the sympathetic and parasympathetic divisions of the autonomic nervous system. Heart Rate Variability (HRV) is measured by using ECG signals. There is a positive association between HRV indices and cognitive performance. 4rth reading will be taken at the time of perturbation along with cognitive loading.
Galvanic Skin Response | Baseline
  Galvanic Skin Response is used in many psychophysiological studies. A change in the electrical property of skin is known as the galvanic skin response. GSR signals are used to capture autonomic nerve responses as a parameter of sweat gland function. There is a direct relation between GSR reading and cognitive loading.
Galvanic Skin Response (2nd reading) | Periprocedural
  Galvanic Skin Response is used in many psychophysiological studies. A change in the electrical property of skin is known as the galvanic skin response. GSR signals are used to capture autonomic nerve responses as a parameter of sweat gland function. There is a direct relation between GSR reading and cognitive loading. 2nd reading will be taken to measure static balance along with cognitive loading.
Galvanic Skin Response (3rd reading) | Periprocedural
  Galvanic Skin Response is used in many psychophysiological studies. A change in the electrical property of skin is known as the galvanic skin response. GSR signals are used to capture autonomic nerve responses as a parameter of sweat gland function. There is a direct relation between GSR reading and cognitive loading. 3rd reading will be taken at the time of perturbation without cognitive loading.
Galvanic Skin Response (4rth reading) | Periprocedural
  Galvanic Skin Response is used in many psychophysiological studies. A change in the electrical property of skin is known as the galvanic skin response. GSR signals are used to capture autonomic nerve responses as a parameter of sweat gland function. There is a direct relation between GSR reading and cognitive loading. 4rth reading will be taken at the time of perturbation along with cognitive loading.
NASA Task Load Index | after static balance with cognitive loading
  The different dimensions of task load, including mental demand, physical demand, temporal demand, performance, effort and frustration, will be measured subjectively using the NASA Task Load Index(TLX). Low ratings will typically indicate an increased cognitive load. 1st reading will be taken after measuring static balance along with cognitive loading.
NASA Task Load Index (2nd reading) | after perturbation with cognitive loading.
  The different dimensions of task load, including mental demand, physical demand, temporal demand, performance, effort and frustration, will be measured subjectively using the NASA Task Load Index(TLX). Low ratings will typically indicate an increased cognitive load. 2nd reading will be taken after perturbation with cognitive loading.

CONTACTS AND LOCATIONS:
Overall Officials: Imran Amjad, PhD, Principal Investigator — Riphah International University
Locations (1):
- Riphah International University, Islamabad, Pakistan

IPD SHARING:
Plan to Share IPD: No